CLINICAL TRIAL: NCT01027221
Title: Randomised Phase I/II Trial in Order to Evaluate the Effect of Neoadjuvant Radiation on Tumor Infiltrating T-cells by Neoadjuvant Low-Dose-Radiation Therapy in Primarily Resectable Pancreatic Cancer
Brief Title: Low Dose Radiation to Improve T-Cell Infiltration in Pancreatic Cancer
Acronym: IMPACT2010
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPACT2010
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2017-11

CONDITIONS: Primarily Resectable Pancreatic Cancer
Keywords: Low Dose Radiation; pancreatic cancer; Immunostimulation
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0 (No Intervention): primarily resectable pancreatic cancer patients
- 0,5 Gy (Active Comparator): neoadjuvant Radiation of 0,5 Gy two days before resection
  Interventions: Radiation: neoadjuvant photon radiation
- 2 Gy (Active Comparator): neoadjuvant Radiation of 2 Gy 2 days before resection
  Interventions: Radiation: neoadjuvant photon radiation
- 5 Gy (Active Comparator): neoadjuvant Radiation of 5 Gy 2 days before resection
  Interventions: Radiation: neoadjuvant photon radiation

INTERVENTIONS:
Radiation: neoadjuvant photon radiation — single fraction, four dimensions (4D) planned, image guided, Radiation at a dose of 0,5 Gy in Intensity modulated radiotherapy (IMRT)-technique 2 days before resection
  Arms: 0,5 Gy
Radiation: neoadjuvant photon radiation — single fraction, 4D-planned, image guided, 2 Gy Radiation to the tumor with a safety margin, in IMRT-technique 2 days before resection
  Arms: 2 Gy
Radiation: neoadjuvant photon radiation — single fraction, 4D-planned, image guided, 5 Gy Radiation to the tumor with a safety margin, in IMRT-technique 2 days before resection
  Arms: 5 Gy

SUMMARY:
Principal purpose of the study is the determination of an active local external beam radiotherapy dose leading to a maximum number of tumor infiltrating T-cells.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis of resectable pancreatic carcinoma is required prior to treatment. Potentially resectable is defined as no extrapancreatic disease, no evidence (on CT) of involvement of the celiac axis or superior mesenteric artery, no evidence (on CT or MRI) of occlusion of the superior mesenteric vein or superior mesenteric-portal venous confluence.
* No evidence of metastatic disease as determined by chest CT scan, abdominal CT scan (or MRI)
* 18 years of age or older
* American Society of Anesthesiologists (ASA)- Performance status of 1 to 3
* Women of child bearing potential must practice adequate contraception and refrain from breast feeding. Female patients must have a negative pregnancy test within 7 days of treatment
* Informed consent

Exclusion Criteria:

* Locally irresectable pancreatic cancer
* distant metastases
* medically unfit for surgery
* Pregnant or lactating women
* prior chemotherapy or radiation treatment
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation
* Unwillingness to participate or inability to comply with the protocol for the duration of the study
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery
* Participation in other interventional trials

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Principal purpose of the study is the determination of an active local external beam radiotherapy dose leading to a maximal number of tumor infiltrating T-cells. The total T-cell activity serves as primary surrogate parameters for anti- tumoral activity | 1 year
  Principal purpose of the study is the determination of an active local external beam radiotherapy dose leading to a maximal number of tumor infiltrating T-cells. The total T-cell activity serves as primary surrogate parameters for anti- tumoral activity

SECONDARY OUTCOMES:
local control and recurrence patterns of pancreatic cancer relative to a standard as seen in historical controls | 5 years
  local control and recurrence patterns of pancreatic cancer relative to a standard as seen in historical controls
surgical morbidity in patients undergoing pancreatic resection who received this protocol treatment | 1 year
  surgical morbidity in patients undergoing pancreatic resection who received this protocol treatment
frequencies of tumor-reactive T-cells in blood and bone marrow | 2 years
  frequencies of tumor-reactive T-cells in blood and bone marrow
expression of migration-relevant adhesion molecules on tumor endothelial cells | 2 years
  expression of migration-relevant adhesion molecules on tumor endothelial cells
expression of proinflammatory cytokines and activation-dependent, immune-associated transcriptionally factors in tumors and blood | 2 years
  expression of proinflammatory cytokines and activation-dependent, immune-associated transcriptionally factors in tumors and blood
quality of life according to the EORTC QoL questionnaire after 6, 12, 18 and 24 months | 3 years
  quality of life according to the EORTC QoL questionnaire after 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter E. Huber, Prof. PhD MD, Principal Investigator — German Cancer Research Centre and Clinic for Radiation Oncology of the University of Heidelberg
Locations (2):
- Germany (2):
  - Clinic for General, Visceral and Transplantation Surgery, Heidelberg
  - German Cancer Research Center, Heidelberg

REFERENCES:
- [Derived] Timke C, Winnenthal HS, Klug F, Roeder FF, Bonertz A, Reissfelder C, Rochet N, Koch M, Tjaden C, Buechler MW, Debus J, Werner J, Beckhove P, Weitz J, Huber PE. Randomized controlled phase I/II study to investigate immune stimulatory effects by low dose radiotherapy in primarily operable pancreatic cancer. BMC Cancer. 2011 Apr 13;11:134. doi: 10.1186/1471-2407-11-134. PMID 21489291